CLINICAL TRIAL: NCT00311142
Title: Actigraphic Sleep Patterns in Newborns Delivered Via Vacuum Extraction vs. Partum Spontaneous and Cesarean Section.
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr. Ayala Maayan, Sheba Medical Center
Other Study IDs: SHEBA-06-3126-AM-CTIL
Record Dates: First submitted 2006-04-04; First posted 2006-04-05 (Estimated); Last update posted 2008-04-16 (Estimated); Status verified 2008-04

CONDITIONS: Healthy
Keywords: Sleep pattern; newborn; actigraphy; delivery mode; Parents' approval

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The development of regular sleep-wake cycle is an important factor of the newborn maturation and it has influence on behavior .Factor that may influence the process of the maturation of the sleep-wake cycle is the delivery mode.nd growing. These various states could be detected and measured with actigraphy, using a wrist-watch like device that continuously measures and records the subject's movements.The present study aims to compare vacuum delivery with regular, elective and not elective caesarean sections. We hypothesize that the sleep of vacuum-delivered newborns will be more fragmented then newborns in other delivery modes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy newborn, born either by regular delivery, vacuum extraction or cesarean section

Exclusion Criteria:

* Preterms, newborns that need special medical treatment and/or repeated blood sampling as glucose.

Ages: 1 Day to 2 Days | Sex: All
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2003-03; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ayala Maayan-Metzger, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Background] Korte J, Hoehn T, Siegmund R. Actigraphic recordings of activity-rest rhythms of neonates born by different delivery modes. Chronobiol Int. 2004 Jan;21(1):95-106. doi: 10.1081/cbi-120027980. PMID 15129826